CLINICAL TRIAL: NCT02153372
Title: Cell Based Therapy by Implanted Bone Marrow-derived Mononuclear Cells (BMC) for Bone Augmentation of Plate-stabilized Proximal Humeral Fractures
Brief Title: Cell Therapy by Bone Marrow-derived Mononuclear Cells (BMC) for Large Bone Defect Repair: Phase-I Clinical Trial
Acronym: BMC2012
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: LOEWE CGT (Unknown)
Responsible Party: Principal Investigator, Ingo Marzi, MD Prof., head physician, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMC2012
Record Dates: First submitted 2014-02-13; First posted 2014-06-03 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Humerus Fracture Displaced Proximal
Keywords: large bone defect, bone marrow-derived mononuclear cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMC2012 (Experimental): The large bone defect was then be bridged as per clinical standard, filled with a clinically established scaffold (ß-TCP), and 1.3 x106/ml BMC were loaded per 1 ml ß-TCP in situ.
  Interventions: Other: BMC2012

INTERVENTIONS:
Other: BMC2012

SUMMARY:
In the present phase-I clinical trial we investigate safety and feasibility of an augmentation with preoperatively isolated autologous BMC cells seeded onto ß-TCP in combination with an angle stable fixation (Philos plate®) for the therapy of proximal humeral fractures.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 50. and 90. years with proximal humerus fractures
* indication for open reposition and internal stabilisation with a proximal fixed- angle plate for humerus (PHILOS, Synthes, Oberdorf, Swiss):
* 2-, 3- or 4-fragment fracture according to NEer
* dislocation of >10 mm between fragments and/or
* angle of > 45° between fragments and/or
* dislocation of tuberculum major > 5 mm
* negative pregnancy test of premenopausal women
* signed informed consent for surgery and participation in the clinical trial

Exclusion Criteria:

* contraindications against administration of Investigational medicinal product (IMP) is pregnancy and nursing
* dislocation fracture
* known psychic disorder that leads to incompliance (e.g. dementia, schizophrenia, major depression)
* pathologic fractures caused by other underlying diseases
* fracture-induced nerve damage
* tumor disease with recent adjuvant therapy or treatment during the last 3 months (e.g. chemotherapy, radiotherapy), untreated tumor diseases
* known hypersensibility against components of the transplant
* participation in a clinical trial during the last 3 months prior to this study

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
safety | at day -1
  Analysis of safety : morbidity of bone marrow punction local reaction (infection, delayed wound healing) systemic reaction (leucocytes, C-reactive protein, Interleukin-6, procalcitonin) fever (> 38,5°C longer than 2 days)
safety | at day 0
  Analysis of safety : morbidity of bone marrow punction local reaction (infection, delayed wound healing) systemic reaction (leucocytes, C-reactive protein, Interleukin-6, procalcitonin) fever (> 38,5°C longer than 2 days)
safety | week 1 post surgery
  Analysis of safety : morbidity of bone marrow punction local reaction (infection, delayed wound healing) systemic reaction (leucocytes, C-reactive protein, Interleukin-6, procalcitonin) fever (> 38,5°C longer than 2 days)
safety | week 6 post surgery
  Analysis of safety : morbidity of bone marrow punction local reaction (infection, delayed wound healing) systemic reaction (leucocytes, C-reactive protein, Interleukin-6, procalcitonin) fever (> 38,5°C longer than 2 days)
safety | week 12 post surgery
  Analysis of safety : morbidity of bone marrow punction local reaction (infection, delayed wound healing) systemic reaction (leucocytes, C-reactive protein, Interleukin-6, procalcitonin) fever (> 38,5°C longer than 2 days)

SECONDARY OUTCOMES:
feasibility | at day-1
  Analysis of feasibility of isolation and application of BMC, logistic and clinical controls
feasibility | at day 0
  Analysis of feasibility of isolation and application of BMC, logistic and clinical controls
feasibility | week 1 post surgery
  Analysis of feasibility of isolation and application of BMC, logistic and clinical controls
feasibility | week 6 post surgery
  Analysis of feasibility of isolation and application of BMC, logistic and clinical controls
feasibility | week 12 post surgery
  Analysis of feasibility of isolation and application of BMC, logistic and clinical controls

OTHER OUTCOMES:
osseous healing by radiologic evaluation | at day 0
  Analysis of fracture healing, consolidation, necrosis, dislocation of reposition, screw cutting
DASH-Score | at 12 weeks post surgery
  testing the function of the shoulder
documentation of concomitant medication and Adverse Events | at day -1
  analysis of medication and Adverse Events
osseous healing by radiologic evaluation | week 1 post surgery
  Analysis of fracture healing, consolidation, necrosis, dislocation of reposition, screw cutting
osseous healing by radiologic evaluation | week 6 post surgery
  Analysis of fracture healing, consolidation, necrosis, dislocation of reposition, screw cutting
osseous healing by radiologic evaluation | week 12 post surgery
  Analysis of fracture healing, consolidation, necrosis, dislocation of reposition, screw cutting
documentation of concomitant medication and Adverse Events | day 0
  analysis of medication and Adverse Events
documentation of concomitant medication and Adverse Events | week 1
  analysis of medication and Adverse Events
documentation of concomitant medication and Adverse Events | week 6 post surgery
  analysis of medication and Adverse Events
documentation of concomitant medication and Adverse Events | week 12 post surgery
  analysis of medication and Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Marzi, MD Prof., Principal Investigator — Department of Trauma-, hand- and reconstructive surgery, Goethe University, Frankfurt
Locations (1):
- Department of trauma-, hand- and reconstructive surgery, Goethe University Hospital, Frankfurt, Theodor-Stern-Kai 7, Germany